CLINICAL TRIAL: NCT04891198
Title: An Open, Single-arm, Multi-center Phase II Clinical Study of ENVAFOLIMAB Single-agent Treatment in Patients With Advanced Solid Tumors
Brief Title: ENVAFOLIMAB Single-agent Treatment in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN035-CN-012
Record Dates: First submitted 2021-04-26; First posted 2021-05-18 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor
Keywords: TMB, solid tumor
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Intervention Model Description: This study is an open, single-arm study, without randomization and blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with TMB-H/TMB-L (Experimental): Subjects receive KN035 400 mg Subcutaneously on Day 1 and day 15 of cycle 1 and on day 1 of every subsequent 4-week cycle (Q4W)
  Interventions: Drug: Envafolimab

INTERVENTIONS:
Drug: Envafolimab — Subcutaneous injection

SUMMARY:
An open, single-arm, multi-center Phase II clinical study of ENVAFOLIMAB single-agent treatment in patients with advanced solid tumors,to compare the overall response rate of TMB-high and TMB-Low,to determine the cut off value between TMB-high and TMB-Low of diagnosis device.Then,observe the efficacy of ENVAFOLIMAB uesd comfirmed TMB-H Value

DETAILED DESCRIPTION:
The enrolled subjects will receive envafolimab treatment during the treatment phase, and the dosage and usage is 400 mg envafolimab subcutaneously injected every four weeks, 28 days as a treatment cycle.

The study treatment continued to reach the standard of stopping treatment. During this period, the efficacy, safety and PK will be evaluated according to the visit process.In this study, imaging examinations (CT or MRI) were used to evaluate the efficacy at baseline and during the study period. The results of the examination were evaluated based on the efficacy evaluation criteria for solid tumors (RECIST1.1) and irRECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate and sign the informed consent form.
2. Age ≥ 18 years old, regardless of gender.
3. Patients with unresectable or metastatic advanced solid tumors confirmed by histology or cytology.
4. Subjects with advanced malignant solid tumors who had disease progression or intolerance and no satisfactory alternative treatment with at least first-line standard treatment.

   Note: If recurrence occurs during adjuvant/neoadjuvant therapy or within 6 months after completion, adjuvant/neoadjuvant therapy is considered to be the first-line treatment for advanced disease.
5. Have not received immune checkpoint inhibitor treatment.
6. Patients with the following tumor types: small cell lung cancer, cervical cancer, endometrial cancer, ovarian cancer, vulvar cancer, neuroendocrine tumors, salivary gland cancer, thyroid papillary or follicular cancer, skin squamous cell carcinoma, skin malignant melanoma , Merkel cell tumor, head and neck squamous cell carcinoma, colorectal cancer, gastric cancer, bladder cancer, cholangiocarcinoma, etc.
7. Have tissue and blood samples that can detect TMB specimen.
8. There is at least one measurable lesion (RECIST 1.1 standard).
9. ECOG score of 0 or 1.
10. The expected survival period is ≥ 12 weeks.
11. Sufficient organ and bone marrow function (no hematopoietic growth factor, blood transfusion or platelet therapy was given within 7 days before the first study drug treatment):

    1. Blood routine: absolute neutrophil count (ANC) ≥1.5×109/L, platelet ≥100×109/L and hemoglobin ≥90 g/L;
    2. Liver function: serum total bilirubin ≤ 1.5 times the upper limit of the normal reference range (×ULN); when there is no liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; ALT and AST ≤5 × ULN in liver metastasis;
    3. Renal function: subjects with serum creatinine ≤ 1.5 × ULN or creatinine level> 1.5 times ULN, measured or calculated according to Cockcroft-Gault formula creatinine clearance rate ≥ 60.0 mL / min;
    4. Coagulation function: International normalized ratio (INR) ≤ 1.5 and partially activated prothrombin time (aPTT) ≤ 1.5 × ULN; (For patients undergoing anticoagulation therapy, the investigator judges that both INR and aPTT are safe and effective treatments Within);
    5. Heart function: left ventricular ejection fraction (LVEF) detected by echocardiography>50%
12. Women with fertility must have a negative serum pregnancy test within 7 days before the first medication. Reproductive male or female patients voluntarily use effective contraceptive methods, such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, intrauterine devices, etc., from signing the informed consent until 90 days after the last study medication. All female patients will be considered fertile unless the female patient has been naturally menopausal, has undergone artificial menopause, or has been sterilized (such as hysterectomy, bilateral adnexectomy).

Exclusion Criteria:

1. Participate in the clinical trials of other investigational drugs or investigational devices within 28 days before the first medication; or have received anti-tumor treatment within 2 weeks, including but not limited to chemotherapy and radiotherapy (allowed to complete the palliative at least 1 week before the study drug treatment Radiotherapy) or targeted therapy.
2. The toxicity of previous anti-tumor treatments has not recovered to 0 or 1 level (hair loss, peripheral neurotoxicity caused by chemotherapy ≤ 2 can be selected). Subjects who need to use corticosteroids (> 10 mg/day prednisone equivalent dose) or other immunosuppressive drugs for systemic therapy within 14 days before the study drug is administered.

   Note: If there is no active autoimmune disease, inhaled or topical steroid hormones, or adrenal hormone replacement therapy with a prednisone equivalent dose of ≤ 10 mg per day is allowed. Allow short-term (≤ 7 days) use of glucocorticoids for preventive treatment (for example, for subjects with a history of severe allergies, when other anti-allergic drugs cannot be used instead to prevent allergy to contrast agents, researchers can use glucocorticoids according to local diagnosis and treatment routines Prevention) or for the treatment of non-autoimmune diseases (for example, delayed type hypersensitivity caused by contact allergens).
3. Subjects who have active, or have had autoimmune diseases or risks that may recur (for example, an organ transplant that requires immunosuppressive therapy). However, subjects with type I diabetes, hypothyroidism requiring only hormone replacement therapy, or skin diseases that do not require systemic treatment (for example, vitiligo, psoriasis, or hair loss) are allowed to be included in the group. For any uncertain situation, it is recommended to consult the sponsor's medical monitor before signing the informed consent.
4. Major surgery (except for biopsy) or the surgical incision did not heal completely within 4 weeks before the first study drug treatment.
5. Suffered from other known malignant tumors within 2 years before enrollment (except for treated skin basal cell carcinoma, skin squamous cell carcinoma and/or carcinoma in situ after radical resection).
6. Untreated brain metastases and Symptomatic brain metastasis or spinal cord compression after treatment ; for patients with brain metastases who have previously received treatment, if the clinical and imaging evidence does not indicate disease progression within 4 weeks before the first study drug treatment, and 2 weeks before the first administration There is no need to receive corticosteroid treatment and can be considered for inclusion.
7. Previous history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia, symptomatic interstitial lung disease or any evidence of active pneumonia detected by chest CT scan within 4 weeks prior to first study drug therapy.
8. Subjects with a history of active tuberculosis infection within 1 year before the first study administration and a history of active tuberculosis infection more than 1 year ago were considered suitable for inclusion if the investigator determined that there was no evidence of active tuberculosis at present.
9. Mental or substance abuse disorders that are known to interfere with test compliance.
10. A history of human immunodeficiency virus (HIV) infection or an active bacterial or fungal infection requiring systematic treatment in the 14 days prior to initial study drug therapy.
11. Uncontrolled hepatitis virus infection (positive for HBV DNA or HCV RNA) .
12. Within 4 weeks of initial administration, there is ascites requiring drainage or diuretic treatment, or pleural or pericardial effusion requiring drainage and/or symptoms of tachypnea.
13. Cardiovascular disease with significant clinical significance.
14. Receive live or attenuated live vaccine within 4 weeks prior to the first study drug treatment.
15. History of severe allergic reaction to humanized antibodies or fusion proteins.
16. Any other disease , and the investigator had reason to suspect that the patient was not eligible for study drug therapy.
17. Part II: The results of tumor tissue samples were MSI-H

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to approximately half past one year
  To evaluate the objective response rate of Envafolimab in patients with advanced solid tumors with high tumor mutation burden (TMB-H) [Blind Independent Imaging Review Committee (BIRC) evaluation]

SECONDARY OUTCOMES:
ORR | Up to approximately half past one year
  To evaluate the objective response rate of Envafolimab in patients with TMB-H and TMB-L advanced solid tumors (investigator assessment)
DCR | Up to approximately half past one year
  To evaluate the disease control rateof Envafolimab in patients with TMB-H and TMB-L advanced solid tumors
DoR | Up to approximately half past one year
  To evaluate the duration of remission of Envafolimab in patients with TMB-H and TMB-L advanced solid tumors
PFS | Up to approximately half past one year
  To evaluate the progression-free survival of Envafolimab in patients with TMB-H and TMB-L advanced solid tumors
OS | Up to approximately half past one year
  To evaluate the overall survival of Envafolimab in patients with TMB-H and TMB-L advanced solid tumors

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided